CLINICAL TRIAL: NCT05621642
Title: The Effect of Telerehabilitation-Based Exercise Training on Breathing, Balance and Gait Parameters in Parkinson's Patients
Brief Title: Telerehabilitation Based Exercise Training in Parkinson's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ilknur Mazı, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-MAZI-001
Record Dates: First submitted 2022-10-28; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Respiration; Gait Disorders, Neurologic
Keywords: telerehabilitation; balance; parkinson
MeSH Terms: conditions — Parkinson Disease; Respiratory Aspiration; Gait Disorders, Neurologic | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Group (Experimental): Trainings will be given to the intervention group patients by the researchers. Respiratory, balance and strengthening exercises suitable for the patients will be applied over an online platform under the supervision of a physiotherapist.
  Interventions: Other: Breathing exercises; Other: Core stabilization exercises; Other: Balance and strengthening exercises
- Offline Group (Active Comparator): The exercises will be video recorded gradually every two weeks and the exercise program of each week will be sent to the patient. The patient will do respiratory, balance and strengthening exercises accompanied by video.
  Interventions: Other: Breathing exercises; Other: Core stabilization exercises; Other: Balance and strengthening exercises

INTERVENTIONS:
Other: Breathing exercises — In the sitting position, the patient does 15 diaphragm breathing and 15 huffing exercises.
Other: Core stabilization exercises — This intervention includes bridging exercise and abdominal exercises.
Other: Balance and strengthening exercises — It includes sitting and standing on the chair 15 times and turning around the chair.

SUMMARY:
Parkinson's disease (PD) is the second most common progressive disease after Alzheimer's disease.It is a progressive, multisystemic and neurodegenerative disease. The prevalence of Parkinson's disease increases with age. increases together. In industrialized countries, people over the age of 60 account for 0.3% of the entire population.It affects about 1% of people and 3% of people over the age of 80 .Patient management with telerehabilitation (TR), chronic heart disease, neurological dysfunction.It is as effective as face-to-face treatment in different clinical conditions such as musculoskeletal and musculoskeletal disorders proven . In addition, TR will increase accessibility and create a less restrictive environment. comparable to traditional rehabilitation as it provides new opportunities to create not only can it be more effective than it . Intense exercise and long-term training In cases where it is necessary, it is accepted to continue exercise therapy with TR programs at home.may be a viable solution.When telerehabilitation-based studies are examined, communication, swallowing and walking are generally focused on parameters. Treatment with telerehabilitation method in PD, Studies investigating the effects on respiratory and postural instability parameters are quite is limited . The aim of this study is to improve telerehabilitation-based exercise training in PD. respiratory muscle strength, cough capacity, dynamic balance, participation in activities of daily living and to investigate its effect on walking parameters. also online physiotherapist.Comparing the effects of supervised exercises and offline video-based exercise training intended.

DETAILED DESCRIPTION:
Parkinson disease (PD) is the most common progressive, multisystemic and neurodegenerative disease after Alzheimer disease. Its prevalence increases with age and rises sharply around the age of 65 . The main pathological change is the progressive degeneration of neurons in the substantia nigra pars compacta, one of the nuclei forming then basal ganglia . Currently, pharmacological treatments are used primarily for symptomatic control and provide only short-term benefits before the disease progresses to a severe stage. Physical activity and exercise can provide cost-effective and universally available aids for current PH treatments. Therefore, it is imperative to examine the effects of exercise on PD. Evidence shows that exercise training is an effective approach to manage symptoms in PD . Physiotherapy interventions in PD aim to maximize functional ability and minimize secondary complications within the scope of patient education and rehabilitation support, and to control unwanted side effects of medical treatment and possible motor fluctuations . Patients who applied to the Neurology Clinic of Bakirkoy Psychiatric and Neurological Diseases Hospital and were diagnosed with idiopathic PH and volunteered to participate in the study will be included in our study. Patients with PD who meet the study inclusion criteria and are between the ages of 50-85 years according to Modified Hoehn & Yahr will be randomly assigned to the intervention and control groups. Patients with PH participating in the study will be randomly assigned to the intervention (Online) and control (Offline) groups. Patients in both groups will participate in a telerehabilitation-based exercise program for 45-60 minutes a day, 3 days a week, for 6 weeks. The intensity of exercise training will be planned to progress gradually every two weeks. In the following weeks, the number of repetitions, the number of sets and the difficulty levels of the exercises will be increased compared to the beginning and the exercises will be continued. Trainings for intervention group patients will be performed by researchers under the supervision of a physiotherapist through an online platform on breathing, balance and strengthening exercises suitable for the patients. For the patients in the control group, the same exercises will be recorded on video every two weeks and the exercise program of each week will be sent to the patient. The patient will be asked to do the exercises accompanied by video. The general evaluation form of the patients and their demographic information, disease history, family history, contact information, education level, and medications will be questioned. Modified Hoehn-Yahr Score and Unified Parkinson Disease Rating Scale (UPDRS) will be used to evaluate disease severity and disability level.Respiratory muscle strength of the patients will be measured using a portable, electronic intraoral pressure measuring device (Carefusion Micromedical, Micro RPM, USA). Peak cough flow will be measured with PEF (peak flow meter).Balance will be evaluated with the Tinetti Balance Scale and the Timed Get Up and Go Test. The 10 m walking test will be used to evaluate walking performance. Participation in activities of daily living and evaluation of patients functional activity status will be performed with the Parkinson Activity Scale . The sample size of the study was calculated with the G*Power 3.1 power analysis program. Considering the effect size of the Timed Up and Go Test, one of the outcome measurements,1.48, the sample size required for 99% working power was calculated at a 95% confidence interval. It was determined that the number of cases to be included for both groups should be at least 19. In order to protect the working power of the cases against the possibility of dropping out of the study, a 10% drop rate will be added to each group and 21 cases will be included . Statistical analysis of the data obtained from the study will be made using the statistical program "Statistical Package for Social Sciences" (SPSS) Version 22.0 (SPSS inc., Chicago, IL, USA). Whether the data are suitable for normal distribution will be determined by the Shapiro-Wilk Test. According to the analysis results of this test, parametric tests will be applied in the analysis of the data that fit the normal distribution, and non-parametric tests will be used in the analysis of the data that do not fit the normal distribution. In the statistical analysis of the study, the evaluated variables will be defined with mean (Mean), standard deviation (SD), confidence interval (CI) and percentage values. Independent Samples T-test for quantitative/numerical data and Chi-squared test for qualitative/non-numerical data will be used to compare the demographic and clinical characteristics of the groups that make up the study. Comparison of the pre-treatment and post-treatment values of the groups will be made with Wilcoxon Signed Rank test or Paired Samples T-test. Comparison of data between groups will be done with Mann Whitney U test or Independent Samples T-test. Effect size of changes within groups, difference between measurements.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with PH by a neurologist,
* Being between 45 and 85 years old,
* Being between I and III according to the modified Hoehn & Yahr Staging (29)
* To have a score of 24 or higher in the Mini Mental State Assessment (30),
* To be taking their medication regularly.

Exclusion Criteria:

* Having an orthopedic disability that will affect balance and mobility,
* Those with serious chronic diseases that will significantly affect their quality of life (congestive heart failure, myocardial infarction),
* Severe dyskinesia, cognitive problem that prevents cooperation,
* Not having internet access with a smart phone or computer,

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-03-13 (Estimated); Study Completion 2023-06-05 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test | 3 minute
  In the timed up and go test, subjects are asked to rise from a standard arm chair, walk to a marker 3 m away, turn, walk back, and sit down again. The test is a reliable and valid test for quantifying functional mobility that may also be useful in following clinical change over time.
Respiratory Strength Assesment | 3 minute
  MIP and MEP value will be measured.
Peak Cough Stream Assesment | 3 minute
  Changed motor control of cough as there is a change in force production using the expiratory muscles

SECONDARY OUTCOMES:
Tinetti balance Test | 5 minute
  To evaluate mobility, balance and gait in the elderly and It has been proposed and widely used to predict falls. It evaluates balance ability and gait under 2 main headings: the first 9 questions are about balance, the next 7 questions are It's about walking. Calculation of the survey score; The total score of the first 9 items gives the balance score, the total score of the next 7 items gives the walking score, and the sum of the balance and walking scores gives the total score. 16 items are the movements made during the activities of daily living. As a result of the evaluation made by observation, it is scored as 0-1-2.
10 m Walking Test | 3 minute
  It is a practical clinical assessment tool developed to measure walking capacity and motor performance of elderly individuals. The 10-meter Walking Test is performed by measuring the time it takes for a person to walk at normal walking speed between two markers that are 10 meters apart .
Parkinson's Activity Scale Parkinson Activity Test | 5 minute
  Parkinson's Activity Scale, a scale developed to evaluate functional activities in PD, provides information about the transfer status of patients. Scored between 0 and 4 points in this scale, a high score indicates good performance. The scale has subsections such as getting up from a chair, in-bed mobilization, and walking akinesia.
Unified Parkinson's Disease Rating Scale | 5 minute
  It will be used to evaluate the severity of the disease and the level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Argün Pulat, Principal Investigator — Doctor in hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee A, Gilbert RM. Epidemiology of Parkinson Disease. Neurol Clin. 2016 Nov;34(4):955-965. doi: 10.1016/j.ncl.2016.06.012. Epub 2016 Aug 18. PMID 27720003
- [Background] Peretti A, Amenta F, Tayebati SK, Nittari G, Mahdi SS. Telerehabilitation: Review of the State-of-the-Art and Areas of Application. JMIR Rehabil Assist Technol. 2017 Jul 21;4(2):e7. doi: 10.2196/rehab.7511. PMID 28733271
- [Background] McCue M, Fairman A, Pramuka M. Enhancing quality of life through telerehabilitation. Phys Med Rehabil Clin N Am. 2010 Feb;21(1):195-205. doi: 10.1016/j.pmr.2009.07.005. PMID 19951786
- [Background] Silverman EP, Sapienza CM, Saleem A, Carmichael C, Davenport PW, Hoffman-Ruddy B, Okun MS. Tutorial on maximum inspiratory and expiratory mouth pressures in individuals with idiopathic Parkinson disease (IPD) and the preliminary results of an expiratory muscle strength training program. NeuroRehabilitation. 2006;21(1):71-9. PMID 16720940
- [Background] Saleem AF, Sapienza CM, Okun MS. Respiratory muscle strength training: treatment and response duration in a patient with early idiopathic Parkinson's disease. NeuroRehabilitation. 2005;20(4):323-33. PMID 16403998
- [Background] Wirdefeldt K, Adami HO, Cole P, Trichopoulos D, Mandel J. Epidemiology and etiology of Parkinson's disease: a review of the evidence. Eur J Epidemiol. 2011 Jun;26 Suppl 1:S1-58. doi: 10.1007/s10654-011-9581-6. Epub 2011 May 28. PMID 21626386
- [Background] Van Den Eeden SK, Tanner CM, Bernstein AL, Fross RD, Leimpeter A, Bloch DA, Nelson LM. Incidence of Parkinson's disease: variation by age, gender, and race/ethnicity. Am J Epidemiol. 2003 Jun 1;157(11):1015-22. doi: 10.1093/aje/kwg068. PMID 12777365
- [Background] Lotankar S, Prabhavalkar KS, Bhatt LK. Biomarkers for Parkinson's Disease: Recent Advancement. Neurosci Bull. 2017 Oct;33(5):585-597. doi: 10.1007/s12264-017-0183-5. Epub 2017 Sep 21. PMID 28936761
- [Background] Kim Y, Lai B, Mehta T, Thirumalai M, Padalabalanarayanan S, Rimmer JH, Motl RW. Exercise Training Guidelines for Multiple Sclerosis, Stroke, and Parkinson Disease: Rapid Review and Synthesis. Am J Phys Med Rehabil. 2019 Jul;98(7):613-621. doi: 10.1097/PHM.0000000000001174. PMID 30844920
- [Background] Cheng DK, Nelson M, Brooks D, Salbach NM. Validation of stroke-specific protocols for the 10-meter walk test and 6-minute walk test conducted using 15-meter and 30-meter walkways. Top Stroke Rehabil. 2020 May;27(4):251-261. doi: 10.1080/10749357.2019.1691815. Epub 2019 Nov 21. PMID 31752634
- [Background] Nieuwboer A, De Weerdt W, Dom R, Bogaerts K, Nuyens G. Development of an activity scale for individuals with advanced Parkinson disease: reliability and "on-off" variability. Phys Ther. 2000 Nov;80(11):1087-96. PMID 11046196
- [Background] Feng H, Li C, Liu J, Wang L, Ma J, Li G, Gan L, Shang X, Wu Z. Virtual Reality Rehabilitation Versus Conventional Physical Therapy for Improving Balance and Gait in Parkinson's Disease Patients: A Randomized Controlled Trial. Med Sci Monit. 2019 Jun 5;25:4186-4192. doi: 10.12659/MSM.916455. PMID 31165721
- [Background] Soke F, Guclu-Gunduz A, Kocer B, Fidan I, Keskinoglu P. Task-oriented circuit training combined with aerobic training improves motor performance and balance in people with Parkinson's Disease. Acta Neurol Belg. 2021 Apr;121(2):535-543. doi: 10.1007/s13760-019-01247-8. Epub 2019 Nov 18. PMID 31741209